CLINICAL TRIAL: NCT02897167
Title: Retrospective and Prospective Study of the Activation of Proinflammatory Pathways of Toll-like Receptors in Patients With Schizophrenia: a Comparative Effect of Risperidone vs Aripiprazole
Brief Title: Study of the Activation of Proinflammatory Pathways of Toll-like Receptors in Schizophrenia Patients
Acronym: PAFIP_TLR
Status: Completed | Type: Observational
Sponsor: Fundación Marques de Valdecilla (Other)
Collaborators: Centro de Investigación Biomédica en Red de Salud Mental (Network); Instituto de Investigación Marqués de Valdecilla (Other)
Responsible Party: Principal Investigator, Benedicto Crespo-Facorro, Professor of Psychiatry, Fundación Marques de Valdecilla
Other Study IDs: PAFIP_TLR
Record Dates: First submitted 2016-09-07; First posted 2016-09-13 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2019-03

CONDITIONS: Schizophrenia; Mental Disorders; Psychotic Disorders
Keywords: Psychosis; Antipsychotic Agents; Immunology; Schizophrenia Spectrum and Other Psychotic Disorders
MeSH Terms: conditions — Schizophrenia; Mental Disorders; Psychotic Disorders; Schizophrenia Spectrum and Other Psychotic Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Serum and peripheral blood mononuclear cell (PBMC)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- PAFIP patients (1): Individuals included in the First Episode Psychosis Clinical Program (PAFIP) between June 2011 and February 2016.
  Retrospective study of frozen samples: samples at baseline and 3 months will be analyzed.
  Interventions: Genetic: Retrospective study of frozen samples
- PAFIP patients (2): Individuals included in the First Episode Psychosis Clinical Program (PAFIP) between September 2016 and September 2017.
  Prospective study of fresh samples: samples at baseline and 3 months will be analyzed.
  Interventions: Genetic: Prospective study of fresh samples
- Controls: Healthy subjects without psychotic disorder.
  Interventions: Genetic: Retrospective study of frozen samples

INTERVENTIONS:
Genetic: Retrospective study of frozen samples — Frozen samples of serum and peripheral blood mononuclear cell (PBMC) stored in the Biobank Valdecilla will be selected.
  Groups: Controls; PAFIP patients (1)
Genetic: Prospective study of fresh samples — Samples of serum and cells will be drawn.
  Groups: PAFIP patients (2)

SUMMARY:
The study of immune pathways involved in the etiopathogeny of schizophrenia would be an important advance to understand the mechanisms involved in the development of this disease and it would be a turning point in drug therapy. Until now, the mechanism of action of antipsychotics focused on the blockade or modulation of brain dopaminergic pathways. If immunological pathways responsible for neuroinflammation and neurodegeneration which involve alterations in different areas and brain pathways (including dopaminergic pathways) are discovered, investigators could develop new treatments that act on these new targets, allowing to delay the onset of the first psychotic episode and improve the evolution and impact of this disease.

DETAILED DESCRIPTION:
Schizophrenia is a mental illness that affects approximately 1% of the population. It supposes an important impact on patients and the socio-health system, since most patients will have difficulty to have an autonomous and independent life and they will need health, economic and social resources for lifetime.

Until recently, the etiopathogeny of schizophrenia was explained by the combination of genetic and environmental factors. However, in recent years there are increasing evidence of the involvement of the immune system in the development and evolution of schizophrenia in at least a subset of patients. Although several meta-analyzes have been published where the increases or decreases in some interleukins and other proinflammatory molecules are described, immune pathways involved in the development and evolution of schizophrenia are still unknown.

The first observations that relate the immune system disorders with the development of non-affective psychosis were made a century ago where it is described the association between pathogen infections (viruses, protozoa or spirochetes) and the occurence of psychosis. Pathogens can directly affect neurons and brain structures, increasing the release of free radicals of oxygen and nitrogen or indirectly altering the activation of the innate or adaptive immune system. They have been published current epidemiological studies that support this theory and they argue that there is an increased risk of having a psychotic decompensation after hospitalization. Furthermore, it is known that many of the genes involved in schizophrenia match those genes involved in the defense against pathogens attack.

Several epidemiological studies have objectified the association of autoimmune diseases and/or chronic inflammatory diseases (intestinal, vasculitis, etc.) with some mental disorders such as schizophrenia, being stress one of the most important triggers factors in the development of both pathologies. Considering that in most cases the onset of autoimmune disease or chronic inflammatory precedes the first psychotic episode, it is hypothesized the autoimmune reaction as a trigger for psychotic symptoms. However, although these studies show statistically significant the involvement of some interleukins (increase in interleukin 6 (IL-6) mainly) in the development or exacerbation of schizophrenia, the levels of interleukins can be altered by other causes such as cardiovascular diseases, obesity and metabolic syndrome; conditions highly prevalent in patients with schizophrenia.

The innate immune system consists of various immune cells (macrophages, mast cells, dendritic cells, microglia, leukocyte, etc.) that recognize pathogen-associated molecular patterns (PAMPs) or damage-associated molecular pattern molecules (DAMPs) through a receptorial system called pattern-recognition receptors (PRRs), located on the cell surface or in cytoplasm. Toll-like receptors (TLRs) are one of the most important families of PRRs. They are transmembrane proteins that have an extracellular domain which binds to the ligands and other intracellular domain which binds to other protein complexes to initiate intracellular transduction pathways. Among the 11 known, the TLRs most studied in schizophrenia has been the TLR-4. Multiple studies have objectified that TLRs are expressed during neurodevelopment in early stages of life and they also have an important role in neurodevelopment and neuronal plasticity during adulthood. Microglia are phagocytic cells located in the central nervous system (CNS) and it is known that they express various types of TLRs. Its role as regulatory cells of CNS is done via intracellular signaling pathways that initiate TLRs. Depending the activated signaling routes, microglia perform different functions: involved positively in the immune response, in neurodevelopmental, in neuronal plasticity and in synaptogenesis, or otherwise through production of proinflammatory cytokines and free radicals of oxygen and nitrogen that favors both neuroinflammation and cerebral neurotoxicity.

Some epidemiological and experimental studies in both animals and humans suggest that infections by viruses, bacteria and protozoa in the prenatal phase (especially in the first quarter) represent a major risk factor for prenatal inflammation, abnormalities in neurodevelopment, obstetric complications and behavioral changes similar to those observed in schizophrenia patients. TLRs can cause neuronal damage in the fetus through two intracellular signaling pathways: increasing cytokine production and/or antimicrobial factors and producing a maintained activation of microglia. Both increased cytokines and antimicrobial factors such as maintained activation of microglia will cause the accumulation of free radicals of oxygen and nitrogen, resulting in neurodegeneration, necrosis and/or apoptosis, which will lead to changes both in the structure and brain function, and in the normal process of child neurodevelopment. It is known that excessive activation of microglia may lead to a reduction in the synapses between glutaminergic neurons in some brain areas such as cerebral cortex, hippocampus and basal ganglia, similar to glutamatergic hypofunction found in brains of schizophrenia patients. In addition, several studies have been published demonstrating the anti-inflammatory and antioxidant properties of antipsychotics, suggesting that its effectiveness is not only due to its action on dopaminergic receptors (classical theory) but they also have a modulatory effect on the immune system.

ELIGIBILITY:
Inclusion Criteria:

* Patients included in the First Episode Psychosis Clinical Program (PAFIP) between June 2011 and September 2017.
* Living in the catchment area.
* Experiencing their first episode of psychosis before 40 years.
* Meeting Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-V) criteria for a principal diagnosis of schizophreniform, schizophrenia, schizoaffective, brief reactive psychosis, or psychosis non otherwise specified.
* No prior treatment with antipsychotic medication or, if previously treated, a total life time of adequate antipsychotic treatment of less than 6 weeks.

Exclusion Criteria:

* Meeting DSM-V criteria for drug dependence.
* Meeting DSM-V criteria for mental retardation.
* Having a history of neurological disease or head injury.

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Individuals included in the First Episode Psychosis Clinical Program (PAFIP) at the University Hospital Marqués de Valdecilla (Santander - Cantabria, Spain) between June 2011 and September 2017.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Measure the expression of proinflammatory molecules of activation pathways of TLRs in patients and controls using the Luminex xMAP technology: a comparative effect of Risperidone vs Aripiprazole. | 3 months
  The Milliplex Human High Sensitivity T Cell Magnetic Bead Kit will be used to analyze the proinflammatory molecules. This kit includes response cytokines (Th1, Th2, Th17 and regulatory) and cytokines secreted by macrophage cells and myeloid lineage. It allows a balance of pro and anti-inflammatory cytokines.
  Luminex is an automated flow cytometer with an open technology that allows various tests to measure different biological parameters, reducing time, handling and cost overruns compared to more traditional methods such as Western Blot, enzyme-linked immunosorbent assay (ELISA) or traditional protein arrays. The methodology uses tests in the microsphere surface or magnetic beads of 5.6 um diameter which emit fluorescence and it is detected in a compact analyzer (Luminex).

SECONDARY OUTCOMES:
Assessment the expression of genes encoding proinflammatory pathways of TLRs in patients and controls using the Luminex xMAP technology. | 3 months
  The Mitogen-Activated and Stress-Activated Protein Kinase (MAPK/SAPK) Signaling Magnetic Bead Kit will be used to detect changes in the lysates of frozen cells of the following proteins: phosphorylated Extracellular Signal-Regulated Kinase (ERK)/MAPK 1/2 (Thr185/Tyr187), STAT1 (Tyr701), Jun Amino-terminal Kinases (JNK) (Thr183/Tyr185), Mitogen-activated protein Kinase kinase 1 (MEK1) (Ser217/221), Mitogen- and Stress-activated protein Kinase 1 (MSK1) (Ser212), Activating Transcription Factor-2 (ATF2) (Thr71), p53 (Ser15), HSP27 (Ser78), c-Jun (Ser73) and p38 (Thr180/Tyr182). This method is a fast and very useful alternative and it is more objective than the Western Blot and conventional immunoprecipitation.
Measure the functionality of proinflammatory pathways of TLRs in patients and controls after direct cell stimulation. | 3 months
  Cells respond to stimuli from the microenvironment by activation of intracellular signaling cascades. Many of these stimuli are transmitted via receptors having in their intracellular domain tyrosine kinases which promote cell metabolism and his growth. Many of these signals activate Ser / Thr kinases signals, whose intermediaries are p70 S6 kinase, MSK1, Signal Transducers and Activators of Transcription (STATs) and Cyclic adenosine monophosphate Response Element-Binding protein (CREB). On the other hand, the danger signals and cell death can promote other signaling pathways such as p38, JNK and p53.

OTHER OUTCOMES:
Compare the long-term evolution of patients with varying degrees of activation of immune system using the Luminex xMAP technology. | 3 years
  To assess whether it can predict the disease progression based on immune activation (quantization the levels of proinflammatory molecules) in the first psychotic episode.

CONTACTS AND LOCATIONS:
Overall Officials: Benedicto Crespo-Facorro, Professor, Principal Investigator — University Hospital Marqués de Valdecilla, IDIVAL, Department of Psychiatry, School of Medicine, University of Cantabria, Santander, Spain. CIBERSAM Centro Investigación Biomédica en Red Salud Mental, Madrid, Spain
Locations (1):
- University Hospital Marqués de Valdecilla, Santander, Cantabria, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pardo-de-Santayana G, Juncal-Ruiz M, Vazquez-Bourgon J, Riesco-Davila L, Ortiz-Garcia de la Foz V, Pelayo-Teran JM, Lopez-Hoyos M, Crespo-Facorro B. Active psychosis and pro-inflammatory cytokines in first-episode of psychosis. J Psychiatr Res. 2021 Feb;134:150-157. doi: 10.1016/j.jpsychires.2020.12.060. Epub 2020 Dec 22. PMID 33385633